CLINICAL TRIAL: NCT05689060
Title: Mulligan Straight Leg Raising Versus Post Facilitation Stretch on Hamstring Flexibility in Physiotherapy Students: Randomized Controlled Trial
Brief Title: Mulligan Straight Leg Raising Versus Post Facilitation Stretch on Hamstring Flexibility in Physiotherapy Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Mahmoud Abd-elmonem, Assist Prof. Physical therapy for pediatric department, faculty of physical therapy , Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mulligan technique
Record Dates: First submitted 2023-01-01; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Rehabilitation
Keywords: mulligan technique; facilitation stretch technique; hamstring; flexibility

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): received mulligan straight leg raising
  Interventions: Other: mulling Straight leg raising technique
- group II (Experimental): received post facilitation stretch on hamstring muscles
  Interventions: Other: post facilitation stretch

INTERVENTIONS:
Other: mulling Straight leg raising technique — Subject was in supine lying, therapist stood at the side of limited, therapist placed subjects flexed knee over therapists shoulder and subject was asked to push therapist away with his leg and then relax. At this point therapist pushed subjects bent knee up as far as in the direction of shoulder.
  Arms: Group I
Other: post facilitation stretch — Muscle energy technique was applied using post facilitation stretch While the participant lying in supine position, the pelvis was strapped down to the table for stabilization and control on accessory movement and the contralateral limb was securely strapped down to the table to prevent excessive hip and pelvic rotations during procedures.The participant's hip was passively flexed and the leg extended until tension was sensed and the participant reported a moderate stretching sensation.
  Arms: group II

SUMMARY:
There are several research on Mulligan's techniques that have demonstrated their effectiveness in lowering hamstring tightness, and Mulligan is a pain-free therapy that may be used on any patients complaining of low back pain and hamstring tightness. the purpose of this preliminary study was to determine the effect of Mulligan technique versus post facilitation stretch technique on hamstring flexibility in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* age 18-25 years
* had 20-50 degrees active knee extension loss with hip and knee in 90 degrees (popliteal angle)

Exclusion Criteria:

* lower limb and spinal deformity,
* hamstring injuries and tightness associated with muscle soreness,
* history of fracture or surgery of back pelvis,

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Active knee extension test | after two months
  Active knee extension test( popliteal angle) is an objective test for measuring tightness of hamstring muscles with electro goniometer while active knee extension. It has been showed excellent inter-rater and intra-rater reliability for assessing hamstring flexibility in asymptomatic healthy adults
Passive compliance | after two months
  Passive compliance is defined as the ratio of change in angle to the change in passive force. A handheld dynamometer (HHD; Micro Manual Muscle Tester; North Coast Medical Inc.) was used to measure the passive torque.

CONTACTS AND LOCATIONS:
Overall Officials: Reham H Diab, Phd, Study Chair — Cairo university, faculty of physical therapy
Locations (1):
- Amira Mahmoud Abd-elmonem, Giza, Egypt